CLINICAL TRIAL: NCT07077070
Title: A Feasibility, Prospective, Repeated-measures, Within-subject, Interventional Study Investigating the Electrical Categorical Loudness Scaling Using the Mobile Research App in the Home and In-clinic Situation in Experienced Adult Cochlear Implant Participants
Brief Title: Investigating Electrical Categorical Loudness Scaling Using a Mobile Research App in Experienced Adult Cochlear Implant Participants
Acronym: ELSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AI5862
Record Dates: First submitted 2025-06-20; First posted 2025-07-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-06

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Cochlear implant; Sensorineural hearing loss; loudness scaling
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Participants receiving both Standard and Fast ELS task (Experimental)
  Interventions: Device: Standard Electrical Categorical Loudness Scaling task (Standard-ELS); Device: Fast Electrical Categorical Loudness Scaling task (Fast-ELS)

INTERVENTIONS:
Device: Standard Electrical Categorical Loudness Scaling task (Standard-ELS) — The Standard-ELS task is conducted using the Mobile Research Application within the Nexus Research system. It is completed in two phases: the first phase identifies the lower and upper bounds of the loudness range based on participant ratings, while the second phase collects data from stimulations delivered within the established range.
Device: Fast Electrical Categorical Loudness Scaling task (Fast-ELS) — The Fast-ELS task employs an algorithm to estimate the lower and upper bounds of the loudness range using a limited number of samples. This range is then refined by collecting additional samples across various loudness categories for comprehensive coverage.

SUMMARY:
This clinical study will evaluate a feature of the investigational Nexus Research System used for programming cochlear implants.

Programming a cochlear implant-commonly referred to as MAP fitting-involves activating the device, allowing recipients to acclimatize to hearing sounds, and then fine-tuning the program based on the user's perception of loudness across different sounds. This process typically occurs over several visits and requires a clinician to collect data for the fine-tuning phase.

The Nexus Research System includes an "Electrical Loudness Scaling" task, which participants can complete independently using a mobile application to collect the necessary data. Based on findings from previous studies, this feature has been revised to enable faster data collection. The current study will assess the performance of the updated feature.

The study will involve experienced cochlear implant users. Participants will use the feature, undergo a series of hearing assessments-including evaluations of loudness perception-and provide feedback on the updated feature.

ELIGIBILITY:
Inclusion Criteria:

* At least three months of experience with the cochlear implant.
* Implanted with the CI600 series (CI612, CI622, CI632) or CI500 series (CI512, CI522, CI532) cochlear implant.
* Able to be programmed with ACE (Advanced Combination Encoder), a fixed pulse width (PW) MAP with a maximum PW of 50 us per channel and with ≥ 18 enabled channels on the sound processor MAP.
* Fluent speaker in the language used to conduct the study procedures, as determined by the investigator.
* Willing and able to provide written informed consent and to comply with all requirements of the protocol.

Exclusion Criteria:

* Participants programmed with an acoustic component in the tested ear.
* Additional health factors, known to the investigator, that would prevent or restrict participation in the evaluations, including significant visual impairment and/or dexterity issues.
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the investigator.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organizations or contractors engaged by Cochlear for the purposes of this investigation.
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless Cochlear sponsored and determined by investigator or Sponsor to not impact this investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-10-21 (Actual); Primary Completion 2025-12-24 (Actual); Study Completion 2025-12-24 (Actual)

PRIMARY OUTCOMES:
Change in patient reported loudness rating scores for very soft sounds (loudness category 5) between Fast-ELS and Standard-ELS within one on-site session. | Day 0, Day 14
  To compare the accuracy of Fast-ELS and Standard-ELS obtained on MRA using a visual analogue scale within one session on-site.
Change in patient reported loudness rating scores for loud sounds (loudness category 35) between Fast-ELS and Standard-ELS within one on-site session. | Day 0, Day 14
  To compare the accuracy of Fast-ELS and Standard-ELS obtained on MRA using a visual analogue scale within one session on-site.
Change in patient reported loudness rating scores for very soft sounds (loudness category 5) between Fast-ELS and Standard-ELS within one at home session. | Day 0 - Day 14
  To compare the accuracy of Fast-ELS and Standard-ELS obtained on MRA using a visual analogue scale within one session at home.
Change in patient reported loudness rating scores for loud sounds (loudness category 35) between Fast-ELS and Standard-ELS within one at home session. | Day 0 - Day 14
  To compare the accuracy of Fast-ELS and Standard-ELS obtained on MRA using a visual analogue scale within one session at home.

SECONDARY OUTCOMES:
Correlation coefficient of very soft sounds (loudness category 5) obtained with Fast-ELS within one session on-site. | Day 0, Day 14
  Test-retest reliability of Fast-ELS outcomes to very soft sounds obtained within one session on-site.
Correlation coefficient of very soft sounds (loudness category 5) obtained with Fast-ELS within one session at home. | Day 0 - Day 14
  Test-retest reliability of Fast-ELS outcomes to very soft sounds obtained within one session at home.
Correlation coefficient of loud sounds (loudness category 35) obtained with Fast-ELS within one session on-site. | Day 0, Day 14
  Test-retest reliability of Fast-ELS outcomes to loud sounds obtained within one session on-site.
Correlation coefficient of loud sounds (loudness category 35) obtained with Fast-ELS within one session at home. | Day 0 - Day 14
  Test-retest reliability of Fast-ELS outcomes to loud sounds obtained within one session at home.
Correlation coefficient of very soft sounds (loudness category 5) obtained with Fast-ELS obtained during multiple sessions on-site. | 14 days
  Test-retest reliability of Fast-ELS outcomes to very soft sounds obtained during multiple sessions on-site.
Correlation coefficient of very soft sounds (loudness category 5) obtained with Fast-ELS obtained during multiple sessions at home. | 14 days
  Test-retest reliability of Fast-ELS outcomes to very soft sounds obtained during multiple sessions at home.
Correlation coefficient of very soft sounds (loudness category 35) obtained with Fast-ELS obtained during multiple sessions on-site. | 14 days
  Test-retest reliability of Fast-ELS outcomes to loud sounds obtained during multiple sessions on-site.
Correlation coefficient of very soft sounds (loudness category 35) obtained with Fast-ELS obtained during multiple sessions at home. | 14 days
  Test-retest reliability of Fast-ELS outcomes to loud sounds obtained during multiple sessions at home.

CONTACTS AND LOCATIONS:
Overall Officials: Anke Plasmans, Study Director — Cochlear Limited
Locations (3):
- Cochlear Denver Research Centre, Lone Tree, Colorado, United States
- Belgium (2):
  - Cochlear Technology Centre Belgium, Mechelen, Mechelen
  - European Institute for Otorhinolaryngology (EIORL), ENT Department, Sint-Augustinus Antwerp, Antwerp

IPD SHARING:
Plan to Share IPD: No